CLINICAL TRIAL: NCT03188887
Title: Treatment of IgA Nephropathy According to Renal Lesions
Acronym: TIGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140931; 2016-004507-31 (EudraCT Number)
Record Dates: First submitted 2017-05-02; First posted 2017-06-16 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: IgA Nephropathy
Keywords: NIgA; Kidney biopsy; GFR; Corticotherapy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Renin-Angiotensin System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): Treatment with Renin Angiotensin system (RAS) blockade or SGLT2i.
  Interventions: Drug: Renin Angiotensin system (RAS) blockade or Inhibitors of sodium glucose transporter 2 (SGLT2i)
- EXPERIMENTAL (Experimental): Corticotherapy + RAS blockade or SGLT2i treatment. Drug injection (intravenous) + tablets
  Interventions: Drug: corticotherapy; Drug: Renin Angiotensin system (RAS) blockade or Inhibitors of sodium glucose transporter 2 (SGLT2i)

INTERVENTIONS:
Drug: corticotherapy — 3 IV pulses steroids followed by oral steroids for 4 months
  Arms: EXPERIMENTAL
Drug: Renin Angiotensin system (RAS) blockade or Inhibitors of sodium glucose transporter 2 (SGLT2i) — treatment with Renin angiotensin system (RAS) blockade or SGLT2i

SUMMARY:
TIGER study (Treatment of IgA nEphropathy according to Renal lesions) is a prospective openly randomized controlled study.

The main objective is to evaluate the efficacy of early corticotherapy + Renin Angiotensin System (RAS) blockade or inhibitors of Sodium glucose transporter 2 (SGLT2i) (versus RAS blockade or SGLT2i alone) after two years of evolution in IgAN patients with severe histological lesions.

DETAILED DESCRIPTION:
Currently, IgAN treatment recommendations are only based on clinico-biological parameters. Steroids therapy appears to have a major role in IgAN treatment, but previous studies evaluating steroids lacked of optimal control group and reproducible evaluation criteria. No prospective study with optimal nephroprotection had included renal pathology in patients selection criteria, although histological evaluation improves patients prognosis prediction. Until now, the lack of a reliable histological classification has precluded the use of histological lesions to evaluate IgAN prognosis and treatment. Given the recently identified major prognostic role of histological lesions in IgAN, we propose to introduce renal pathology to guide the treatment of IgAN in a multicenter study, using currently validated evaluation criteria of chronic kidney disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Patient with IgAN
3. Renal biopsy < 45 days before inclusion visit
4. PCR ratio >0.75 g/g (within 30 days before or after the renal biopsy)
5. Renal biopsy with at least 8 glomeruli, disclosing at least 2 criteria among:

   * mesangial proliferation (according to Oxford criteria)
   * endocapillary proliferation (according to Oxford criteria)
   * tubulointerstitial fibrosis (according to Oxford criteria) >25% of the biopsy
   * segmental glomerulosclerosis (according to Oxford criteria)
   * at least 1 cellular/fibrocellular crescents (C1 according to Oxford criteria)
6. Patient with Social Security Insurance or CMU
7. Patient having signed an informed consent

Exclusion Criteria:

1. >30% increase of serum creatinine after starting nephroprotection therapy (≥ 15 days and ≤ 6 weeks) only for patient under nephroprotection <45 days of the inclusion visit
2. >50% cellular/fibrocellular crescents, or >50% tubulointerstitial fibrosis or >50% globally sclerotic glomeruli
3. Nephrotic syndrome with minimal change disease and IgA deposits
4. eGFR <20 ml/min/1,73m2 (CKD-EPI formula) within 30 days before or after the renal biopsy
5. Uncontrolled blood pressure (Systolic blood pressure >180 mmHg or diastolic blood pressure > 110 mmHg)
6. Previous corticosteroids treatment (>20 mg/d during more than 15 days, within the last 3 months before the renal biopsy)
7. Pregnancy or breast feeding or women without sufficient contraception
8. Secondary known forms of IgAN
9. Henoch-Schoenlein purpura
10. Additional other chronic renal disease
11. Contraindication for immunosuppressive therapy, including active intestinal bleeding, active gastric or duodenal ulcer; active infection; any malignancy in a last years before the inclusion; severe psychiatric disease; living vaccines; anti-inflammatory dosages of acetylsalicylic acid
12. Contraindication for RAS orSGLT2i blockade therapy
13. Known allergy or intolerance to corticoids or lactose
14. Organ transplant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Failure at 24 months | Month 24
  Failure at 24 months will be defined as :
  * Proteinuria/creatinuria ratio (PCR) > 0,5 g/g
  * or mGFR < 80% of initial mGFR (or eGFR if unavailable)
  * or loss of more than 10 ml/min/1,73m2 of initial mGFR (or eGFR if unavailable)
  * or end stage renal disease (ESRD)
  * or renal transplantation
  * or death

SECONDARY OUTCOMES:
Failure at 6 months | Month 6
  Failure at 6 months will be defined as:
  * PCR > 0.75 g/g
  * or PCR > 0.5 g/g and >30% of initial PCR
  * or eGFR < 80% of initial eGFR
  * or end stage renal disease (ESRD)
  * or renal transplantation
  * or death
Failure at 12 months | Month 12
  Failure at 12 months will be defined as:
  * PCR > 0.75 g/g
  * or PCR > 0.5 g/g and > 30% of initial PCR
  * or mGFR < 80% of initial mGFR (or eGFR if unavailable)
  * or end stage renal disease (ESRD)
  * or renal transplantation
  * or death
Proportion of patients with persistent severe histological lesions in repeat kidney biopsy at 12 months | Month 12
  to compare the evolution of histological lesions between treatment groups at 12 months
Evolution of GFR at 12 months assessed as :- the absolute value of GFR - the absolute difference of GFR from the baseline - the annual degradation (ml/min /1,73m2/year) of GFR during the 12 months | Month 12
  to compare the evolution of measured GFR (mGFR) between treatment groups at 12 months (or estimated GFR (eGFR) if unavailable)
Evolution of GFR at 24 months assessed as :- the absolute value of GFR - the absolute difference of GFR from the baseline - the annual degradation (ml/min /1,73m2/year) of GFR during the 24 months | Month 24
  to compare the evolution of measured GFR (mGFR) between treatment groups at 24 months (or estimated GFR (eGFR) if unavailable)
Evolution of proteinuria assessed as : - the absolute value of proteinuria at 12 and 24 months - the absolute difference of proteinuria from baseline at 12 and 24 months | Month 12 and 24
  to compare the evolution of proteinuria in each group
SF36 scale at 12 months | Month 12
  to compare the quality of life in each therapeutic group
SF36 scale at 24 months | Month 24
  to compare the quality of life in each therapeutic group
Number of side effects | Month 24
  to assess the tolerance of treatments in each therapeutic group
Prognosis markers of failure at 24 months | Month 24
  Clinical, histological, and biological data (including PCR ratio, eGFR and mGFR, renal histological lesions) will be compared between patients with or without failure.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique JOLY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Eric ALAMARTINE, Principal Investigator — CHU SAINT-ETIENNE; Khalil El Karoui, Study Chair — Henri Mondor University Hospital
Locations (1):
- Hôpital Necker Enfants-malades, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi S, Roberts ISD, Wang Z, Jiang L, Tang C, Wang J, Lv J, Wong MG, Barbour SJ, Perkovic V, Cattran D, Zhang H; TESTING Study Pathology Group. Predictive Value of the Oxford Classification for the Effect of Glucocorticoid Therapy in IgA Nephropathy. J Am Soc Nephrol. 2026 Jan 1;37(1):150-159. doi: 10.1681/ASN.0000000796. Epub 2025 Jul 8. PMID 40627446
- [Derived] El Karoui K, Fervenza FC, De Vriese AS. Treatment of IgA Nephropathy: A Rapidly Evolving Field. J Am Soc Nephrol. 2024 Jan 1;35(1):103-116. doi: 10.1681/ASN.0000000000000242. Epub 2023 Sep 29. PMID 37772889